CLINICAL TRIAL: NCT03055754
Title: Endoscopic Argon Plasma Coagulation Vs. Observation In The Management Of Weight Regain After Gastric Bypass Surgery: A Randomized Controlled Trial
Brief Title: Endoscopic Argon Plasma Coagulation Vs. Control For Weight Regain After Gastric Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Clinic and Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KaiserCH
Record Dates: First submitted 2017-01-30; First posted 2017-02-16 (Actual); Last update posted 2019-05-29 (Actual); Status verified 2019-05

CONDITIONS: Obesity; Weight Gain
MeSH Terms: conditions — Obesity; Weight Gain

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Argon randomized arm (Experimental): Endoscopic procedure with a full inventory, measurement of the anastomosis diameter, and an argon plasma coagulation. Followup of all patients by a multidisciplinary team (life, food orientations).
  Interventions: Procedure: Argon randomized arm
- Control arm (Active Comparator): Full inventory and measurement of the anastomosis diameter, without any intervention. Followup of all patients by a multidisciplinary team (life, food orientations).
  Interventions: Procedure: Control arm

INTERVENTIONS:
Procedure: Argon randomized arm — Endoscopic argon plasma coagulation
  Arms: Argon randomized arm
Procedure: Control arm — No Endoscopic procedure
  Arms: Control arm

SUMMARY:
Bariatric surgery procedures have consistently been demonstrated to reduce long-term co-morbidities and mortality. Despite its benefits, weight regain is common, usually initiating around two years after the initial procedure, the underlying mechanism often being an enlargement of the anastomosis diameter for the Roux-en-Y gastric bypass. Although a reduction in the anastomosis diameter has been reported in association with endoscopic argon plasma coagulation, to our knowledge this therapy has not been formally tested in a randomized controlled trial. the objective of this study is to conduct a randomized, parallel controlled trial comparing endoscopic argon plasma coagulation to reduce the enlargement of the anastomosis diameter for the Roux-en-Y gastric bypass versus control with an initial diagnostic endoscopic followed by observation. The investigators hypothesize that the argon coagulation arm will achieve greater weight reduction, with a low incidence of adverse events.

DETAILED DESCRIPTION:
This will be a parallel randomized controlled trial with a 1:1 allocation ratio, comparing endoscopic argon plasma coagulation to reduce the enlargement of the anastomosis diameter for the Roux-en-Y gastric bypass versus control with an initial diagnostic endoscopic followed by observation. The study is designed and reported in accordance with the CONSORT statement for parallel randomized trials. Eventual changes made to the design after trial commencement will be fully reported, including changes in eligibility criteria throughout the study.

Ethical aspects: The study will undergo full review by the local Institutional Review Board, all potential participants being provided with informed consent. Study protocol will only be initiated after consent is signed.

Participants: Inclusion criteria will involve all consecutive patients who have previously undergone a bariatric procedure and who now present with symptoms of weight regain, difficulty maintaining weight, and lack of satiety after meals. The investigator will not exclude any patients meeting these criteria. No other treatments will be provided. A total of 40 participants will be part of this analysis, or 20 per randomization arm.

Setting: Data will be collected at the Kaiser Clinic in São José do Rio Preto, Brazil. Participant accrual will start in April of 2016, with the end of follow-up occurring around the end of 2017.

Interventions: Interventions for the argon randomized arm will include an endoscopic procedure with a full inventory, measurement of the anastomosis diameter, and an argon plasma coagulation. The control arm will only undergo a full inventory and measurement of the anastomosis diameter, without any intervention. Participants allocated to the observational arm and presenting with continued symptoms of weight regain, difficulty maintaining weight, and lack of satiety after meals will not be prevented from undergoing an argon intervention, although our analyses will still analyze their results within the observation arm, thus observing an intention to treat protocol.

Outcomes: Primary outcomes of interested will be weight regain, gastrointestinal symptoms, and satiety verbal analog scale. Secondary outcome measures will include fasting glucose concentration, HbA1c concentration, body weight, body mass index, waist circumference, arterial blood pressure, plasma total cholesterol, HDL cholesterol and triglycerides, quality of life, surgical complications, and diabetes-related complications.

Sample size: The sample size is estimated to be 40 participants total, or 20 in each randomization arm.

Randomization: The random sequence will be generated using the statistical language R by a researcher not involved with subject allocation. The randomization schedule has a blocking size of an undisclosed size, with no stratification. Randomization will be implemented by an administrative assistant using sealed, sequentially numbered envelopes. Researchers will be specifically instructed not to attempt to break the randomization schedule in any manner. Subject allocation will be performed by the principal investigator (GQ) soon after consent and prior to the endoscopic procedure. Given the nature of this intervention, the only individual blinded regarding randomization will be the data analyst. Blinding will be ensured by having codes in the final dataset.

ELIGIBILITY:
Inclusion Criteria:

* all consecutive patients who have previously undergone a bariatric procedure
* who present with symptoms of weight regain, difficulty maintaining weight, and lack of satiety after meals.

Exclusion Criteria:

-

Ages: 16 Years to 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2016-05; Primary Completion 2017-02 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
Weight regain | 48 weeks

SECONDARY OUTCOMES:
Gastrointestinal symptoms | 48 weeks
  Symptoms like Nausea, Vomiting, Cramps in stomach
Satiety verbal analog scale | 48 weeks
Fasting glucose concentration in mg/dL | 48 weeks
HbA1c in percentage | 48 weeks
Arterial blood pressure in mm Hg | 48 weeks
plasma total cholesterol, HDL cholesterol and triglycerides (mg/dL) | 48 weeks
Quality of life of patient | 48 weeks
  Quality of life measured using EQ-5D scale
Surgical and diabetes-related complications | 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Luiz G de Quadros, MD, Principal Investigator — Kaiser Clinic and Hospital
Locations (1):
- Kaiser Clinic and Day Hospital, São José do Rio Preto, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Schulz KF, Altman DG, Moher D; CONSORT Group. CONSORT 2010 statement: updated guidelines for reporting parallel group randomized trials. Obstet Gynecol. 2010 May;115(5):1063-1070. doi: 10.1097/AOG.0b013e3181d9d421. No abstract available. PMID 20410783